CLINICAL TRIAL: NCT02462538
Title: A "Window of Opportunity" Trial With Brentuximab Vedotin and Imatinib in Patients With Relapsed or Refractory ALK+ Anaplastic Large Cell Lymphoma or Patients Ineligible for Chemotherapy
Brief Title: Brentuximab Vedotin and Imatinib in Patients With Relapsed or Refractory ALK+ ALCL
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Due to slow recruitment, recruitment of new patients was stopped, FU was completed for enrolled patients
Sponsor: Arbeitsgemeinschaft medikamentoese Tumortherapie (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AGMT_ALCL1
Record Dates: First submitted 2015-05-18; First posted 2015-06-04 (Estimated); Last update posted 2022-03-03 (Actual); Status verified 2022-02

CONDITIONS: ALK+ Anaplastic Large Cell Lymphoma
MeSH Terms: interventions — Brentuximab Vedotin; Imatinib Mesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Brentuximab vedotin and Imatinib (Experimental): Brentuximab vedotin (every 3 weeks i.v., 1.8 mg/kg) and imatinib (200mg daily orally, escalated from 100mg daily) for up to 48 weeks
  Interventions: Drug: Brentuximab vedotin; Drug: Imatinib

INTERVENTIONS:
Drug: Brentuximab vedotin — Brentuximab vedotin is given in a 21 day cycle intravenously starting at 1.8 mg/kg on day 1 of the first cycle and will be administered by IV infusion given over approximately 30 minutes on day 1 of each 21-day cycle.
  Other Names: Adcetris
Drug: Imatinib — Imatinib will be given orally at a dose of 100mg daily starting from day 1 of the first cycle. The dose will be increased to 200mg daily starting from day 1 of the second cycle if no DLT occurs during the first cycle and will be continued at 200mg for 48 weeks.
  Other Names: Glivec

SUMMARY:
This is an open label pilot study of combining BV in a licensed indication with imatinib in patients with ALCL. It is intended as a "window of opportunity" trial in which the study drugs will be given as an initial substitute for conventional chemotherapy with the intention to achieve a remission enabling the patients to proceed to autologous or allogeneic stem cell transplantation, if eligible.

DETAILED DESCRIPTION:
Patients will be included in this trial if they have relapsed or refractory ALK+ ALCL after at least one line of conventional chemotherapy or if they are ineligible for conventional chemotherapy.

Imatinib will be given continuously starting from day 1 of the first cycle at an oral dose of 100mg daily. The dose will be increased to 200mg daily starting from day 1 of the second cycle if no DLT occurs during the first cycle. BV will be given 3 weekly starting on day 1 at a dose of 1.8 mg/kg body weight. In the absence of a dose limiting toxicity (DLT) i.e. haematological toxicity ≥ grade 2, non- haematological toxicity ≥ grade 3, after 3 weeks of therapy, and in the presence of a clinical response (CR or PR) after cycle 1, the BV dose will continue every 3 weeks for 48 weeks. Dose modifications and stopping rules will be introduced as described in chapter 6. In case of progression at any time during the study the patient will go off trial and receive salvage treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years of age
* ALK+ ALCL
* Histologically confirmed relapse after having achieved a PR or CR with conventional therapy
* Refractoriness to conventional chemotherapy (SD or PD after conventional chemotherapy)
* Not able to receive conventional chemotherapy (e.g. due to comorbidities)
* Adequate organ function, defined as the following:

  * Absolute neutrophil count ≥ 1,500/μL unless there is known hematologic/solid tumor marrow involvement
  * Platelet count ≥ 75,000/ μL unless there is known marrow involvement of the disease
  * Total bilirubin must be < 1.5 x the upper limit of the normal (ULN) unless the elevation is known to be due to Gilbert syndrome.
  * ALT or AST must be < 3 x the upper limit of the normal range. AST and ALT may be elevated up to 5 times the ULN if their elevation can be reasonably ascribed to the presence of hematologic/solid tumor in liver.
  * Serum creatinine must be < 2.0 mg/dL and/or creatinine clearance or calculated creatinine clearance > 40 mL/minute.
  * Hemoglobin must be ≥ 8g/dL.
* Written, voluntarily signed informed consent
* Female patient is either post-menopausal for at least 1 year before the screening visit or surgically sterile or if of childbearing potential, must practice 2 effective methods of contraception, at the same time, from the time of signing the informed consent until 6 months after the last doses of BV and until last doses of imatinib, whatever occurs later, or agrees to completely abstain from heterosexual intercourse.
* Male patients, even if surgically sterilized, (i.e., status post vasectomy) agree to practice effective barrier contraception during the entire study period and through 6 months after the last dose of BV, or agrees to completely abstain from heterosexual intercourse.

Exclusion Criteria:

* Patient has received any other investigational treatment within 28 days before study entry
* Known hypersensitivity to recombinant proteins, murine proteins, or to any excipient contained in the drug formulation of brentuximab vedotin or imatinib
* ECOG performance status ≥ 3
* Acute or chronic infections
* Female patients who are pregnant or breast-feeding
* Known diagnosis of HIV
* Known hepatitis B surface antigen-positive, or known or suspected active hepatitis C infection
* Any serious medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with the completion of treatment according to the protocol.
* Known cerebral or meningeal disease (HL or any other etiology), including signs or symptoms of PML
* Symptomatic neurologic disease compromising normal activities of daily living or requiring medications
* Any sensory or motor peripheral neuropathy greater than or equal to Grade 2
* Known history of any of the following cardiovascular conditions

  * Myocardial infarction within 2 years of study entry
  * New York Heart Association (NYHA) Class III or IV heart failure
  * Evidence of current uncontrolled cardiovascular conditions, including cardiac arrhythmias, congestive heart failure (CHF), angina, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities
  * Recent evidence (within 6 months before first dose of study drug) of a left-ventricular ejection fraction <50%
* Any active systemic viral, bacterial, or fungal infection requiring systemic antibiotics within 2 weeks prior to first study drug dose
* Diagnosed or treated for another malignancy within 3 years before the first dose or previously diagnosed with another malignancy and have evidence of residual disease. Patients with nonmelanoma skin cancer or carcinoma in situ of any type are not excluded if they have undergone complete resection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2015-11-03 (Actual); Primary Completion 2021-11-03 (Actual); Study Completion 2021-11-03 (Actual)

PRIMARY OUTCOMES:
Safety of brentuximab vedotin and imatinib regime as measured by type, frequency and severity of adverse events (AEs) and their relationship to study treatment | up to 6 years

SECONDARY OUTCOMES:
Efficacy of brentuximab vedotin and imatinib regime as measured by proportion of patients responding to treatment | up to 6 years
Ability to receive further Treatment as measured by number of patients being able to receive transplantation | up to 6 years
Progression-free survival as measured by proportion of patients displaying progressive disease | up to 6 years
Overall survival as measured by documentation of deaths | up to 6 years

CONTACTS AND LOCATIONS:
Overall Officials: Ulrich Jäger, MD, Principal Investigator — Universitätsklinik für Innere Medizin I: Klinische Abteilung für Hämatologie und Hämostaseologie
Locations (1):
- Universitätsklinik f. Innere Medizin I, AKH Wien, Klinische Abteilung für Hämatologie und Hämostaseologie, Vienna, Austria